CLINICAL TRIAL: NCT04682782
Title: Intraoperative Small-dose Esketamine Infusion for Pain Control in Burn Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020-516
Record Dates: First submitted 2020-12-03; First posted 2020-12-24 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: Burns
MeSH Terms: conditions — Burns | interventions — Esketamine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Esketamine (Experimental): Participants randomized to this arm will receive Esketamine (1 mg/ml) infused at 0.1 mg/kg/hour (0.1 ml/kg/h) throughout the operation
  Interventions: Drug: Esketamine
- Saline (Placebo Comparator): Participants randomized to this arm will receive 0.9 mg/ml sodium chloride, infused at a rate of 0.1 ml/kg/hour throughout the operation
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Esketamine — Esketamine is infused through the whole period of surgery. Participants randomized to the esketamine arm will receive 1 mg/ml solution infused at 0.1 mg/kg/hour (0.1 ml/kg/h) .
  Arms: Esketamine
Drug: Saline — Participants randomized to the placebo arm will receive 0.9 mg/ml sodium chloride, infused at a rate of 0.1 ml/kg/hour throughout the surgery.
  Other Names: Placebo
  Arms: Saline

SUMMARY:
This study aim to determine whether a small-dose esketamine infusion can be used for pain control in severe burn patients, and thereby reduce the total intra-operative opioid requirement. Secondary objectives are to determine whether this low-dose esketamine infusion will increase the stability of circulation.

ELIGIBILITY:
Inclusion Criteria:

* All intubated adult burn patients( age>18 ), presenting to the operating room;
* Burn area> 30%.

Exclusion Criteria:

* Allergy to Esketamine or benzodiazepines
* Esketamine or ketamine use in the preceding 24 hours
* Increased intracranial pressure
* Increased intraocular pressure
* Porphyria
* Thyroid disorders
* Seizures
* Acute myocardial ischemia
* Children (patients under age 18), prisoners, pregnant or breastfeeding women, patients with psychosis, patients with developmental delay, and any condition which, in the opinion of the investigator, would prevent full participation in this study or would interfere with the evaluation of the trial endpoints.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2020-07-14 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Intraoperative sufentanil | 24 hours
  For all participants, the dose of intraoperative sufentanil will be recorded in micrograms and compared between the two arms.

SECONDARY OUTCOMES:
Intraoperative blood pressure | 24 hours
  For all participants, blood pressure will be recorded and compared between the two arms.
Intraoperative heart rate | 24 hours
  For all participants, heart rate will be recorded and compared between the two arms.
Intraoperative cardiac index | 24 hours
  For all participants, cardiac index will be recorded and compared between the two arms.
Post-operative recovery time | 24 hours
  For all participants, the recovery time of spontaneous breathing will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Min YAN, MD, Principal Investigator — 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China
Locations (1):
- 2nd affiliated hospital, School of Medicine, Zhejiang Universtiy, China, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No